CLINICAL TRIAL: NCT06949501
Title: The Effectiveness of Virtual Patient Simulation Versus Peer Simulation in Enhancing Attitudes, Beliefs, and Skills in Providing Sexual Counseling During Pregnancy
Brief Title: The Effectiveness of Virtual Patient Simulation Versus Peer Simulation in Providing Sexual Counseling During Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Principal Investigator, NESLİHAN YILMAZ SEZER, ASSOCIATE PROFESSOR, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03.03.2025/05-87
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy; Sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual patient simulation group (Experimental)
  Interventions: Other: virtual patient simulation
- peer simulation conducted in a virtual environment group (Experimental)
  Interventions: Other: peer simulation conducted in a virtual environment
- face-to-face peer simulation group (Experimental)
  Interventions: Other: face-to-face peer simulation

INTERVENTIONS:
Other: virtual patient simulation — Students in this group are expected to provide sexual counseling to a virtual patient model following theoretical training. In this context, a virtual patient model has been developed with whom the students will engage for the counseling process.
  Arms: virtual patient simulation group
Other: peer simulation conducted in a virtual environment — Students in this group are expected to provide sexual counseling to their peers in a virtual environment following theoretical training. In the virtual peer simulation, students will see the same background displayed in the virtual patient simulation; however, instead of interacting with a virtual patient, they will connect with a peer via an online platform to conduct the counseling session.
  Arms: peer simulation conducted in a virtual environment group
Other: face-to-face peer simulation — Students in this group are expected to provide sexual counseling to their peers following theoretical training. In the peer simulation, students will conduct their sessions in a communication skills laboratory designed to resemble a clinical consultation room.
  Arms: face-to-face peer simulation group

SUMMARY:
The aim of this study is to compare, in a multidimensional manner, the effectiveness of different educational methods-virtual patient simulation and peer simulation-in improving sexual counseling skills during pregnancy among nursing faculty students.

The study will evaluate three different training methods: virtual patient simulation, peer simulation conducted in a virtual environment, and face-to-face peer simulation. To determine the effectiveness of peer simulation and virtual patient simulation in sexual health counseling, multimodal data collection and analysis methods will be used. These methods will contribute to the development of counseling skills by examining in detail the verbal and non-verbal communication elements exhibited by participants during their interactions with virtual patients and peers. Throughout the research process, students' demographic characteristics, sexual attitudes and beliefs, sexual counseling skills, learning satisfaction and self-confidence levels, opinions on system usability, eye-tracking data, and body movements will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to provide care for pregnant women - Providing informed consent to participate in the study

Exclusion Criteria:

* Having suspended enrollment or taken a leave of absence from education.
* Having received formal education aimed at developing sexual counseling skills.
* Wearing glasses (as it may interfere with the use of wearable eye-tracking systems).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Sexual Attitudes and Beliefs | immediately before the training-immediately after the training
  Students' sexual attitudes and beliefs will be assessed using the the sexual attitudes and belief survey. This scale is a six-point Likert-type scale, with scores ranging from a minimum of 12 to a maximum of 72. Higher scores indicate more negative attitudes and beliefs toward sexual care.
Learning Satisfaction and Self-Confidence | immediately after the training
  Learning satisfaction and self-confidence will be measured using the Student Satisfaction and Self-Confidence in Learning Scale. This scale is a five-point Likert-type scale, with responses ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores reflect greater student satisfaction and self-confidence in learning.
Sexual Counseling Skills | During simulation
  Students' sexual counseling skills will be assessed using the Sexual Counseling Skills Assessment Form. This form is developed based on the BETTER, PLISSIT, Ex-PLISSIT, and One-to-One models, and it covers the entire counseling process from initiation to conclusion. Each item is scored as 0 (not demonstrated) or 1 (demonstrated). The total score ranges from 0 to 34, with higher scores indicating a higher level of skill. The form will be completed while students simulate their counseling skills.
System Usability Opinions | immediately after the training
  Students' opinions regarding system usability will be assessed using the System Usability Scale (SUS). The SUS is a 10-item instrument scored on a five-point Likert scale. Scores range from a minimum of 10 to a maximum of 100. Higher scores indicate higher perceived usability of the system.
Eye Tracking | During simulation
  Eye tracking parameters in the study will be assessed using a wearable eye-tracking system. This device will analyze the areas of focus during students' interactions with virtual patients and peers. The analysis of gaze points and eye movements will help evaluate the distribution of attention during communication.
Body Movements | During simulation
  Body movements will be evaluated using a motion tracking device. These motion detection systems will analyze body language to assess participants' capacity to establish effective connections with virtual patients and peers. This method aims to evaluate participants' ability to use gestures and body language effectively to build strong relationships with patients.

IPD SHARING:
Plan to Share IPD: No